CLINICAL TRIAL: NCT04431063
Title: Comparison of the Functional Outcome of Site Peroneus Longus Graft Donors With and Without Distal Stump Suturing of Peroneus Tendon Brevis on ACL Reconstruction Case .
Brief Title: Comparison of the Functional Outcome of Site Peroneus Longus Graft Donors With and Without Distal Stump Suturing of Peroneus Tendon Brevis on ACL Reconstruction Case in Cipto Mangunkusumo Hospital in Jakarta With 24 Patient as Subject Who Will Divide Into 2 Group.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andri Maruli Tua Lubis, Orthopaedic Surgeon, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-10-1173
Record Dates: First submitted 2020-06-03; First posted 2020-06-16 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: ACL; Rupture of ACL; Donor site; Peroneus Longus Graft; Distal Stump; Peroneus Brevis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sutured Stump (Experimental): The group consist of subject with distal stump suturing of perobeus longus agains peroneus brevis in ACL Reconstruction Case
  Interventions: Procedure: Distal Stump Suturing
- Unsutured Stump (No Intervention): The group consist of subject without distal stump suturing of peroneus longus agains peroneus brevis in ACL Reconstruction Case

INTERVENTIONS:
Procedure: Distal Stump Suturing — in ACL Reconstruction case , Group A consist of subject with operation procedure suturing the distal stump peroneus longus against the peroneus brevis in ACL reconstruction using the peroneus longus autograft.
  Arms: Sutured Stump

SUMMARY:
Injury of the Anterior Cruciate Ligament (ACL) is one of the most common sports injuries. The incidence rate reaches 68.6 cases per 100,000 people per year. Management of ACL injuries for individuals who want to return to the level of exercise activity as before, mostly in the form of reconstructive surgery. As many as 60,000 to 175,000 cases of ACL reconstruction per year are carried out in the United States At present, many reconstructive surgeries are performed by taking tendon grafts on the patient's own body (autograft) to then be used instead of the ACL. The most widely used graft sources are Hamstring and Bone-Patellar Tendon-Bone (BPTB) grafts. Other alternative grafts are Quadriceps tendon, Fascia Lata, Iliotibial Band, and Peroneus Longus Tendon. Each graft retrieval technique has advantages and disadvantages. BPTB graft has the best tensile strength and bone union with bone, but the complications of anterior knee pain are also quite common (5-55%). Hamstring grafts and Quadriceps grafts minimize the complications of anterior knee pain, with fairly good tensile strength, but the union of grafts with bone takes longer. The loss of Hamstring tendons also causes a decrease in muscle strength in Hamstring, where Hamstring has an important role in preventing the anterior translation of the tibia Peroneus Longus Tendon graft is an alternative graft developed to minimize complications associated with graft use from the area around the knee. Peroneus Longus tendons also have tensile strength similar to Hamstring tendons.

As with other graft extracts, Peroneus Longus tendon graft is also accompanied by complications in the donor site. Possible complications arising from the loss of the Peroneus Longus tendon include ankle instability and decreased flexion strength of the 1st ray and ankle eversion. Research carried out by Bancha et al showed a reduction in flexion strength of 1st ray and ankle eversion significantly, without any instability in the ankle. Peroneus longus provides 5.5% strength for moderate dorsiflexion for ankle eversion movements, peroneus longus is the main muscle. But in other studies it is said that the use of peroneus longus graft does not interfere with the stability of the ankle and ROM. Does not even affect the functional outcome of the ankle However, in a study conducted by Bancha et al and Kerimoglu et al., The technique used for taking Peroneus Longus graft tendons did not include suturing in the distal stump of Peroneous Longus. So with this study, researchers wanted to find out whether different results would be found related to donor site complications if the technique used included suturing the distal stump of the Peroneus Longus tendon against the peroneus brevis tendon

ELIGIBILITY:
Inclusion Criteria:

* Patients with total ACL rupture using peroneus longus graft
* The suturing procedure for the distal stump peroneus longus against the peroneus brevis tendon is performed by orthopedic specialists or resident chiefs who have been given training in advance.

Exclusion Criteria:

* Osteoarthtis Knee Kellgren-Lawrence III and IV
* Osteoarthtis Knee Kellgren-Lawrence III and IV
* Flatfoot as evidenced by physical examination and footprinting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Preoperative hand dynamometer value | This measurement was carried out at the preoperative setting
  Value of objective measurement of the strength of the medial part of the plantarflexion in the one metatarsal head with the hand of the Dynamometer when the patient is supine. The measurement is done 3 times and the value used is the average of the 3 times the measurement. Healthy ankles were also examined as a comparison with the same measurement method. There is no minimum and maximum value, and the higher value the better the outcome
Three-months postoperative hand dynamometer value | This measurement was carried out at 3 months postoperatively
  Value of objective measurement of the strength of the medial part of the plantarflexion in the one metatarsal head with the hand of the Dynamometer when the patient is supine. The measurement is done 3 times and the value used is the average of the 3 times the measurement. Healthy ankles were also examined as a comparison with the same measurement method. There is no minimum and maximum value, and the higher value the better the outcome
Six-months postoperative hand dynamometer value | This measurement was carried out at 6 months postoperatively
  Value of objective measurement of the strength of the medial part of the plantarflexion in the one metatarsal head with the hand of the Dynamometer when the patient is supine. The measurement is done 3 times and the value used is the average of the 3 times the measurement. Healthy ankles were also examined as a comparison with the same measurement method. There is no minimum and maximum value, and the higher value the better the outcome
Preoperative Clark's Angle Value | This measurement was carried out at the preoperative setting
  the value of the objective angle measurement on the footprint by drawing a line from the medial side of the one metatarsal head and the heel against the second line which is connecting the one metatrsal head and the peak of the medial longitudinal arch. Clarke Angle of < 31° means there is tendency to flatness and/or pronation. angle of 31° to < 45° is the normal range. Clarke Angle of > 45° means there is tendency to cavus foot
Three-months Clark's Angle Value | This measurement was carried out at the 3 months postoperatively
  the value of the objective angle measurement on the footprint by drawing a line from the medial side of the one metatarsal head and the heel against the second line which is connecting the one metatrsal head and the peak of the medial longitudinal arch. Clarke Angle of < 31° means there is tendency to flatness and/or pronation. angle of 31° to < 45° is the normal range. Clarke Angle of > 45° means there is tendency to cavus foot
Six-months Clark's Angle Value | This measurement was carried out at the 6 months postoperatively
  the value of the objective angle measurement on the footprint by drawing a line from the medial side of the one metatarsal head and the heel against the second line which is connecting the one metatrsal head and the peak of the medial longitudinal arch. Clarke Angle of < 31° means there is tendency to flatness and/or pronation. angle of 31° to < 45° is the normal range. Clarke Angle of > 45° means there is tendency to cavus foot
Preoperative the American Orthopedic Foot and Ankle Score (AOFAS) | Examination carried out 4 times for each patient in preoperative setting
  the questionnaire for assessing the function of both injured feet and ankles and the knee that is in the process of healing. AOFAS score has the range of value of 0 to 100. 0 is the worst value and 100 is the best value possible
Three months postoperative the American Orthopedic Foot and Ankle Score (AOFAS) | Examination carried out 4 times for each patient in 3 months postoperatively
  the questionnaire for assessing the function of both injured feet and ankles and the knee that is in the process of healing. AOFAS score has the range of value of 0 to 100. 0 is the worst value and 100 is the best value possible
Six months postoperative the American Orthopedic Foot and Ankle Score (AOFAS) | Examination carried out 4 times for each patient in 6 months postoperatively
  the questionnaire for assessing the function of both injured feet and ankles and the knee that is in the process of healing. AOFAS score has the range of value of 0 to 100. 0 is the worst value and 100 is the best value possible
Preoperative visual analogue scale foot and ankle (VAS-FA) | Examination carried out 4 times for each patient at preoperative setting
  the questionnaire for assessing the function of both injured feet and ankles and the knee that is in the process of healing. VAS-FA score has the range of value of 0 to 100. 0 is the worst value and 100 is the best value possible
Three-months postoperative visual analogue scale foot and ankle (VAS-FA) | Examination carried out 4 times for each patient at 3 months postoperatively
  the questionnaire for assessing the function of both injured feet and ankles and the knee that is in the process of healing. AS-FA score has the range of value of 0 to 100. 0 is the worst value and 100 is the best value possible
Six-months postoperative visual analogue scale foot and ankle (VAS-FA) | Examination carried out 4 times for each patient at 6 months postoperatively
  the questionnaire for assessing the function of both injured feet and ankles and the knee that is in the process of healing. AS-FA score has the range of value of 0 to 100. 0 is the worst value and 100 is the best value possible

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lyman S, Koulouvaris P, Sherman S, Do H, Mandl LA, Marx RG. Epidemiology of anterior cruciate ligament reconstruction: trends, readmissions, and subsequent knee surgery. J Bone Joint Surg Am. 2009 Oct;91(10):2321-8. doi: 10.2106/JBJS.H.00539. PMID 19797565
- [Background] Angthong C, Chernchujit B, Apivatgaroon A, Chaijenkit K, Nualon P, Suchao-in K. The Anterior Cruciate Ligament Reconstruction with the Peroneus Longus Tendon: A Biomechanical and Clinical Evaluation of the Donor Ankle Morbidity. J Med Assoc Thai. 2015 Jun;98(6):555-60. PMID 26219159
- [Background] Cerulli G, Placella G, Sebastiani E, Tei MM, Speziali A, Manfreda F. ACL Reconstruction: Choosing the Graft. Joints. 2013 Jun 12;1(1):18-24. eCollection 2013 Mar. PMID 25606507
- [Background] Kerimoglu S, Aynaci O, Saracoglu M, Aydin H, Turhan AU. [Anterior cruciate ligament reconstruction with the peroneus longus tendon]. Acta Orthop Traumatol Turc. 2008 Jan-Feb;42(1):38-43. doi: 10.3944/aott.2008.038. Turkish. PMID 18354276
- [Background] Silver RL, de la Garza J, Rang M. The myth of muscle balance. A study of relative strengths and excursions of normal muscles about the foot and ankle. J Bone Joint Surg Br. 1985 May;67(3):432-7. doi: 10.1302/0301-620X.67B3.3997956.
- [Background] Frobell RB, Roos EM, Roos HP, Ranstam J, Lohmander LS. A randomized trial of treatment for acute anterior cruciate ligament tears. N Engl J Med. 2010 Jul 22;363(4):331-42. doi: 10.1056/NEJMoa0907797. PMID 20660401
- [Background] Mentiplay BF, Perraton LG, Bower KJ, Adair B, Pua YH, Williams GP, McGaw R, Clark RA. Assessment of Lower Limb Muscle Strength and Power Using Hand-Held and Fixed Dynamometry: A Reliability and Validity Study. PLoS One. 2015 Oct 28;10(10):e0140822. doi: 10.1371/journal.pone.0140822. eCollection 2015. PMID 26509265
- [Background] Click Fenter P, Bellew JW, Pitts T, Kay R. A comparison of 3 hand-held dynamometers used to measure hip abduction strength. J Strength Cond Res. 2003 Aug;17(3):531-5. doi: 10.1519/1533-4287(2003)0172.0.co;2. PMID 12930182
- [Background] Surburg PR, Suomi R, Poppy WK. Validity and reliability of a hand-held dynamometer with two populations. J Orthop Sports Phys Ther. 1992;16(5):229-34. doi: 10.2519/jospt.1992.16.5.229. PMID 18796754
- [Background] Murley GS, Tan JM, Edwards RM, De Luca J, Munteanu SE, Cook JL. Foot posture is associated with morphometry of the peroneus longus muscle, tibialis anterior tendon, and Achilles tendon. Scand J Med Sci Sports. 2014 Jun;24(3):535-41. doi: 10.1111/sms.12025. Epub 2013 Jan 10. PMID 23301865
- [Background] Pita-Fernandez S, Gonzalez-Martin C, Seoane-Pillado T, Lopez-Calvino B, Pertega-Diaz S, Gil-Guillen V. Validity of footprint analysis to determine flatfoot using clinical diagnosis as the gold standard in a random sample aged 40 years and older. J Epidemiol. 2015;25(2):148-54. doi: 10.2188/jea.JE20140082. Epub 2014 Nov 8. PMID 25382154
- [Background] Gonzalez-Martin C, Pita-Fernandez S, Seoane-Pillado T, Lopez-Calvino B, Pertega-Diaz S, Gil-Guillen V. Variability between Clarke's angle and Chippaux-Smirak index for the diagnosis of flat feet. Colomb Med (Cali). 2017 Mar 30;48(1):25-31. PMID 28559643
- [Background] Quatman CE, Hewett TE. The anterior cruciate ligament injury controversy: is "valgus collapse" a sex-specific mechanism? Br J Sports Med. 2009 May;43(5):328-35. doi: 10.1136/bjsm.2009.059139. Epub 2009 Apr 15. PMID 19372087
- [Background] McGuine TA, Winterstein AP, Carr K, Hetzel S. Changes in Health-Related Quality of Life and Knee Function After Knee Injury in Young Female Athletes. Orthop J Sports Med. 2014 Apr 22;2(4):2325967114530988. doi: 10.1177/2325967114530988. eCollection 2014 Apr. PMID 26535324
- [Background] Beynnon BD, Johnson RJ, Abate JA, Fleming BC, Nichols CE. Treatment of anterior cruciate ligament injuries, part I. Am J Sports Med. 2005 Oct;33(10):1579-602. doi: 10.1177/0363546505279913. PMID 16199611
- [Background] Beynnon BD, Johnson RJ, Abate JA, Fleming BC, Nichols CE. Treatment of anterior cruciate ligament injuries, part 2. Am J Sports Med. 2005 Nov;33(11):1751-67. doi: 10.1177/0363546505279922. PMID 16230470
- [Background] Mihelic R, Jurdana H, Jotanovic Z, Madjarevic T, Tudor A. Long-term results of anterior cruciate ligament reconstruction: a comparison with non-operative treatment with a follow-up of 17-20 years. Int Orthop. 2011 Jul;35(7):1093-7. doi: 10.1007/s00264-011-1206-x. Epub 2011 Feb 2. PMID 21287172
- [Background] Schindler OS. Surgery for anterior cruciate ligament deficiency: a historical perspective. Knee Surg Sports Traumatol Arthrosc. 2012 Jan;20(1):5-47. doi: 10.1007/s00167-011-1756-x. Epub 2011 Nov 22. PMID 22105976
- [Background] Felmet G. Implant-free press-fit fixation for bone-patellar tendon-bone ACL reconstruction: 10-year results. Arch Orthop Trauma Surg. 2010 Aug;130(8):985-92. doi: 10.1007/s00402-010-1050-2. Epub 2010 Jan 22. PMID 20094723
- [Background] Willis-Owen CA, Hearn TC, Keene GC, Costi JJ. Biomechanical testing of implant free wedge shaped bone block fixation for bone patellar tendon bone anterior cruciate ligament reconstruction in a bovine model. J Orthop Surg Res. 2010 Sep 2;5:66. doi: 10.1186/1749-799X-5-66. PMID 20813059
- [Background] Pavlik A, Hidas P, Tallay A, Toman J, Berkes I. Femoral press-fit fixation technique in anterior cruciate ligament reconstruction using bone-patellar tendon-bone graft: a prospective clinical evaluation of 285 patients. Am J Sports Med. 2006 Feb;34(2):220-5. doi: 10.1177/0363546505279920. Epub 2005 Oct 6. PMID 16210575
- [Background] Dargel J, Schmidt-Wiethoff R, Schneider T, Bruggemann GP, Koebke J. Biomechanical testing of quadriceps tendon-patellar bone grafts: an alternative graft source for press-fit anterior cruciate ligament reconstruction? Arch Orthop Trauma Surg. 2006 May;126(4):265-70. doi: 10.1007/s00402-005-0048-7. Epub 2005 Sep 17. PMID 16172862
- [Background] van Eck CF, Kropf EJ, Romanowski JR, Lesniak BP, Tranovich MJ, van Dijk CN, Fu FH. Factors that influence the intra-articular rupture pattern of the ACL graft following single-bundle reconstruction. Knee Surg Sports Traumatol Arthrosc. 2011 Aug;19(8):1243-8. doi: 10.1007/s00167-011-1427-y. Epub 2011 Feb 11. PMID 21311861
- [Background] Zaffagnini S, Marcacci M, Lo Presti M, Giordano G, Iacono F, Neri MP. Prospective and randomized evaluation of ACL reconstruction with three techniques: a clinical and radiographic evaluation at 5 years follow-up. Knee Surg Sports Traumatol Arthrosc. 2006 Nov;14(11):1060-9. doi: 10.1007/s00167-006-0130-x. Epub 2006 Aug 15. PMID 16909301
- [Background] Mohtadi NG, Chan DS, Dainty KN, Whelan DB. Patellar tendon versus hamstring tendon autograft for anterior cruciate ligament rupture in adults. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD005960. doi: 10.1002/14651858.CD005960.pub2. PMID 21901700
- [Background] Freedman KB, D'Amato MJ, Nedeff DD, Kaz A, Bach BR Jr. Arthroscopic anterior cruciate ligament reconstruction: a metaanalysis comparing patellar tendon and hamstring tendon autografts. Am J Sports Med. 2003 Jan-Feb;31(1):2-11. doi: 10.1177/03635465030310011501. PMID 12531750
- [Background] Lee YH, Kuroda R, Zhao J, Chan KM. A tale of 10 European centres - 2010 APOSSM travelling fellowship review in ACL surgery. Sports Med Arthrosc Rehabil Ther Technol. 2012 Jul 28;4(1):27. doi: 10.1186/1758-2555-4-27. PMID 22839644
- [Background] van Dijk PA, Lubberts B, Verheul C, DiGiovanni CW, Kerkhoffs GM. Rehabilitation after surgical treatment of peroneal tendon tears and ruptures. Knee Surg Sports Traumatol Arthrosc. 2016 Apr;24(4):1165-74. doi: 10.1007/s00167-015-3944-6. Epub 2016 Jan 23. PMID 26803783
- [Background] Lin TW, Cardenas L, Soslowsky LJ. Biomechanics of tendon injury and repair. J Biomech. 2004 Jun;37(6):865-77. doi: 10.1016/j.jbiomech.2003.11.005. PMID 15111074
- [Background] Yang G, Rothrauff BB, Tuan RS. Tendon and ligament regeneration and repair: clinical relevance and developmental paradigm. Birth Defects Res C Embryo Today. 2013 Sep;99(3):203-222. doi: 10.1002/bdrc.21041. PMID 24078497
- [Result] Sanders TL, Maradit Kremers H, Bryan AJ, Larson DR, Dahm DL, Levy BA, Stuart MJ, Krych AJ. Incidence of Anterior Cruciate Ligament Tears and Reconstruction: A 21-Year Population-Based Study. Am J Sports Med. 2016 Jun;44(6):1502-7. doi: 10.1177/0363546516629944. Epub 2016 Feb 26. PMID 26920430